CLINICAL TRIAL: NCT06150274
Title: Simplifying Percutaneous Balloon Mitral Valvulotomy (PBMV) to Reduce the Burden of Mitral Stenosis in Sub-Saharan Africa.
Brief Title: Comparison of Wire Assisted Percutaneous Balloon Mitral Valvulotomy With Standard Inoue Balloon Valvulotomy
Acronym: CROSSVal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 523036
Record Dates: First submitted 2023-11-07; First posted 2023-11-29 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2023-11

CONDITIONS: Rheumatic Heart Disease
MeSH Terms: conditions — Rheumatic Heart Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- standard Inoue balloon technique (Active Comparator): Those randomized to the standard care will undergo the procedure using the contemporary Inoue balloon system (Toray Industries, Japan), which is available in 4 sizes: 24, 26, 28 and 30 mm.
  Interventions: Device: Percutaneous Balloon Mitral Valvulotomy
- wire assisted crossing (Active Comparator): The procedure is performed on a similar fashion until atrial septal entry. Once the atrial wall is traversed, and the Mullins sheath is within the left atrium, the mitral valve is crossed with a flexible 0.032- or 0.035 in- 145 cm J-tipped wire. This step could be assisted by a steerable sheath. Once the mitral valve is crossed, the initial wire will be exchanged with a looped stiff wire (Safari or similar) to the left ventricle by use of a 5/6 f pigtail catheter. A commercially available balloon is used to perform the valvulotomy/commissurotomy procedure. Choice of balloon size is made following the formula: Balloon size = patient height (cm)/10 + 10. Fine tuning of the balloon size will be performed peri-operative based on transesophageal echo findings. Use of a separate stiff wire placed in the left atrium/pulmonary vein to ease passage through the atrial septum is left to the discretion of the operator based on the anatomical challenges faced during the procedure.
  Interventions: Device: Percutaneous Balloon Mitral Valvulotomy

INTERVENTIONS:
Device: Percutaneous Balloon Mitral Valvulotomy — Stenotic mitral valve will be dilated to open the commissures

SUMMARY:
The goal of this randomised study is comparison of wire assisted balloon mitral valvulotomy to standard Inoue balloon technique on patients with rheumatic mitral stenosis. The main question it aims to answer is whether procedure time is reduced using the wire assisted method. Participants will be randomized to one of the two methods.

DETAILED DESCRIPTION:
Background: Rheumatic valvular disease, a chronic sequela of acute rheumatic fever, is a leading cause of cardiovascular mortality in developing countries. The available options of management include surgical treatment and balloon valvulotomy. Among various forms of rheumatic valvular lesions, severe mitral stenosis with favorable morphology can be successfully treated by balloon valvulotomy.

Methods: The study is a randomized controlled trial with intervention in both arms.

The objective of this study is to compare procedural time as a primary end point.

ELIGIBILITY:
Inclusion Criteria:

* significant mitral stenosis
* low Wilkins score (< 10)
* mitral regurgitation grade not more than 2

Exclusion Criteria:

* high Wilkins score (>10)
* unfavourable anatomy
* presence of left appendage thrombus
* non-conclusive periprocedural trans oesophageal echocardiography imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Reduction in procedure duration | day 1
  procedure time in minutes

SECONDARY OUTCOMES:
procedure failure | day 1
  failed procedure after lengthy attempt

OTHER OUTCOMES:
mortality | 30 days
  short and long term survival
mortality | 3 months
  short and long term survival
Hospitalization for heart failure | 2 year
  hospitalization for worsening heart failure
Procedure related neurological events | day 1
  new neurological events
Procedure related neurological events | 30 days
  new neurological events
Vascular complications requiring intervention | day 1
  transfusion requiring bleeding or vascular complication requiring percutaneous or surgical intervention
new arrythmia | day 1
  previously non existing arrythmia registered after intervention
new bradyarrythmia | day 1
  new bradyarrythmia requiring device intervention

CONTACTS AND LOCATIONS:
Overall Officials: Nigussie Bogale, MD, PhD, Principal Investigator — Haukeland University Hospital, Bergen, Norway
Locations (1):
- Tikur Anbessa Specialized Hospital, Addis Ababa, Addis Abeba, Ethiopia

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: November 2023 through december 2026
Access Criteria: application must be submitted and signed electronically. The study team will asess the submitted proposals.
URL: http://www.helse-bergen.no